CLINICAL TRIAL: NCT07077707
Title: A Randomized Trial of Chatbot for Prenatal Genetic Counseling
Brief Title: Prenatal Genetics Chatbot Trial: Prenatal GENEie
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melissa Russo, Assistant Professor, Maternal Fetal-Medicine & Genetics, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2164485; R01HD111426 (NIH)
Record Dates: First submitted 2025-02-28; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Genetic Counseling
Keywords: prenatal genetics; prenatal testing; mobile application; chatbot; patient education; aneuploidy; decisional conflict; genetics health literacy
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person genetic counseling (Active Comparator): Patients in this group will be scheduled for an in-person genetic counseling visit to discuss options for aneuploidy screening, carrier screening, and prenatal diagnosis. For Spanish-speaking patients the genetic counselors will use in-person interpreters.
  Interventions: Other: In-person genetic counseling
- Prenatal Genetics Chatbot- Prenatal GENEie (Experimental): Patients in the intervention group will be assisted by research staff to download and interact with the chatbot Prenatal GENEie in their preferred language (English or Spanish) for a minimum of 30 minutes to learn about aneuploidy screening, carrier screening and prenatal diagnosis.
  Interventions: Other: Prenatal GENEie Chatbot

INTERVENTIONS:
Other: Prenatal GENEie Chatbot — Patient Educational Phone Chatbot Application for Prenatal Genetics in English & Spanish
  Arms: Prenatal Genetics Chatbot- Prenatal GENEie
Other: In-person genetic counseling — Standard in-person genetic counseling for prenatal genetics education
  Arms: In-person genetic counseling

SUMMARY:
During pregnancy, all pregnant people are offered tests to look for genetic conditions in the baby. However, there isn't a standard way of giving this information to patients. Doctors have a lot of things to discuss during the first prenatal visit and don't always have time to explain genetics in detail. Also, not everyone has access to genetic counselors. Prenatal genetics can be confusing, especially for people who haven't had a lot of formal education or who speak languages other than English. There might be misunderstandings about what these tests can find and what their benefits or risks are for these tests.

Mobile apps, like chatbots, could be a helpful way to give information about prenatal genetics. Almost everyone has a cell phone, and a chatbot can let people learn at their own speed and whenever they want.

The goal of this study is to see if a chatbot app Prenatal GENEie can teach pregnant women about prenatal genetics, and compare the chatbot to talking with a genetic counselor in person. The study wants to answer these main questions:

* Does the Prenatal GENEie help pregnant patients learn about prenatal genetics the same way as a meeting with a genetic counselor?
* Can the Prenatal GENEie and in-person counseling both help people make decisions about whether they want prenatal genetic testing?

The researchers will compare the chatbot Prenatal GENEie with in-person counseling to see if the chatbot teaches people about prenatal genetics in a similar way.

Participants will:

* Take a test to check what they already know about prenatal genetics prior to the intervention
* Use the chatbot or have an in-person meeting with a genetic counselor
* Take a test after using the chatbot or meeting with a counselor to see how much their knowledge has improved
* Fill out a survey about how comfortable they feel with their decision to do or not do prenatal genetic testing

DETAILED DESCRIPTION:
Current recommendations from the American College of Obstetricians and Gynecologists (ACOG) call for all pregnant people to be offered screening and diagnostic testing options for aneuploidy, including maternal serum screening, cell-free fetal DNA (cfDNA), chorionic villus sampling, amniocentesis, and carrier screening for cystic fibrosis and spinal muscular atrophy. As a result, the nearly 4 million pregnant people receiving prenatal care in the United States annually require access to associated, and complex, prenatal genetic counseling. Additionally, access to pregnancy terminations has radically changed in the post-Dobbs era. With these considerations and a commitment to person centered-care, informed decision-making is critical, and predicated on people having adequate knowledge of the benefits and risks of different testing options. In the context of prenatal genetics, no option is the correct choice for all persons. Instead, the ideal choice is based on an individual's beliefs and values. Obstetric care providers have the challenge of addressing an ever-increasing number of topics during the first prenatal care visit, and prenatal genetic counselors face a high number of referrals. Yet there is a national shortage of genetic counselors with an uneven geographic distribution. The resulting lack of access to standardized prenatal genetic counseling can lead to patient misinterpretation of the goals or results of prenatal genetic testing and may be contributing to socioeconomic and racial disparities in prenatal genetic screening and diagnosis. Minority patients have a lower uptake of prenatal genetic screening and higher live-birth rates of children with Down syndrome likely due to lower rates of informed choice rather than negative attitudes about testing. Language barriers further exacerbate misunderstanding of prenatal genetic testing options.

Mobile digital tools, including chatbots, provide an attractive alternative to in-person genetic counseling due to the near ubiquitous availability of mobile devices among patients and ability to ensure tailoring and standardization. Previous digital tools developed for prenatal genetic education showed promise, but most are more instructional than interactive, computer-based rather than mobile-based, and do not include information on carrier screening currently recommended by ACOG. Notably, most tools were developed before the clinical availability of cfDNA testing, now the most common prenatal screening modality in the U.S. To address this critical need, a multidisciplinary team of perinatologists, genetic counselors, and digital health experts developed an innovative, patient-informed, mobile chatbot (iPrenatal) to simulate a text and audio-based counseling discussion about aneuploidy screening and diagnosis . Preliminary data from the researchers' randomized trial of 258 English-speaking pregnant people showed significantly higher post-intervention knowledge scores among patients who used iPrenatal compared with those who received routine provider education (66% vs 55%, p < 0.001). The researchers propose to leverage this success by engaging users in formative work to create Prenatal GENEie, with information on aneuploidy and carrier testing, and provide all content in English and Spanish. The researchers will evaluate Prenatal GENEie in a randomized controlled trial of 1470 pregnant people in clinics serving racially and socioeconomically diverse pregnant women. The researchers will test their central hypothesis that an enhanced digital education chatbot providing standardized yet tailored prenatal genetic counseling will be comparable to in-person prenatal counseling by a genetic counselor in increasing patient knowledge and uptake of prenatal genetic tests.

The specific aims of this study are:

Aim 1: Determine the effect of Prenatal GENEie on patient knowledge and uptake of prenatal genetic testing, compared to in-person genetic counseling. The researchers hypothesize that Prenatal GENEie will result in non-inferior knowledge gain and testing uptake, compared to genetic counseling.

Aim 2: Assess ability of Prenatal GENEie to narrow the gap in knowledge and uptake of prenatal genetic screening between English- and Spanish-speaking patients, compared to in-person genetic counseling. The researchers hypothesize that Prenatal GENEie will narrow the gap in knowledge scores and uptake of prenatal genetic testing between English- and Spanish-speaking patients.

The expected outcome of this study is high-quality evidence on the ability of an educational chatbot to equitably increase patient knowledge and uptake of prenatal genetic screening and diagnostic tests. If shown to be effective, this validated chatbot interface will be adaptable and scalable to other settings, including areas of provider shortages, and languages to increase equitable access to prenatal genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking with ability to read and write
* Gestational age <20 weeks
* Access to smartphone or tablet (through personal use or study)

Exclusion Criteria:

* Patients who have already had genetic counseling related to current pregnancy
* h/o trisomy, major fetal anomaly. or aneuploidy in previous pregnancy
* Parent with Robertsonian translocation
* Twins, vanishing twin, multi-gestation pregnancy
* Fetal anomaly noted in early pregnancy
* In- vitro fertilization with pre-implantation genetic testing (PGT-A or PGT-M)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1470 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Prenatal Knowledge Score | Baseline knowledge at enrollment and within 7 days after intervention
  The prenatal knowledge score is calculated from questionnaire with 30 true/false questions. The scores range from 0 (lowest knowledge) to 30 (highest knowledge), reflecting the number of correct responses.. The change in prenatal knowledge score is then calculated from the percent answered correctly after the intervention from number of correct responses before the intervention. The highest knowledge increase is 30 and the lowest is 0.
Rate of Prenatal Screening | Assessed between enrollment and 24 weeks gestation
  Proportion of patients who have had cfDNA screening during pregnancy

SECONDARY OUTCOMES:
Rate of Any Prenatal Screening or Diagnostic Testing | Assessed between enrollment and 24 weeks gestation
  Proportion of patients who have any kind of genetic testing: cfDNA, serum screening, carrier screening, diagnostic testing
Decisional-conflict scale | Within 7 days after intervention
  The Decisional-conflict scale consists of 10 items, each with 3 response categories (yes, no, unsure). Items are given a score value of (0=yes, 2=unsure, 4=no). Total score is calculated by summing items, dividing by 10 and multiplying by 25. Score ranges from 0 (no conflict) to 100 (highest decisional conflict) with higher scores indicating higher level of decisional conflict.
Satisfaction Scale for Educational Intervention | Within 7 days after intervention
  Likert Scale for Satisfaction with genetic counseling or chatbot (secondary outcomes to be described in secondary manuscripts). The Likert scale is 1 to 5 with 1= not at all satisfied with the educational intervention to 5=highly satisfied with educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Method Tuuli, MD, Principal Investigator — Women & Infants Hospital in Providence RI
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocols, and metadata including participant age, sex, race and ethnicity, height, weight, socioeconomic status, and other demographic data; past and present medical, surgical and obstetric history; intervention, chatbot genetic counseling or in person genetic counseling; and pregnancy and study outcomes data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2029 in perpetuity
Access Criteria: Data will be findable for the research community. All publications will be made available via the NIH publication policy. Each of the datasets will have an assigned digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.

REFERENCES:
- [Background] Larion S, Warsof SL, Romary L, Mlynarczyk M, Peleg D, Abuhamad AZ. Uptake of noninvasive prenatal testing at a large academic referral center. Am J Obstet Gynecol. 2014 Dec;211(6):651.e1-7. doi: 10.1016/j.ajog.2014.06.038. Epub 2014 Jun 19. PMID 24954652
- [Background] Carlson LM, Harris S, Hardisty EE, Hocutt G, Vargo D, Campbell E, Davis E, Gilmore K, Vora NL. Use of a novel computerized decision aid for aneuploidy screening: a randomized controlled trial. Genet Med. 2019 Apr;21(4):923-929. doi: 10.1038/s41436-018-0283-2. Epub 2018 Sep 14. PMID 30214066
- [Background] Rothwell E, Johnson E, Wong B, Rose NC, Latendresse G, Altizer R, Zagal J, Smid M, Watson A, Botkin JR. The Use of a Game-Based Decision Aid to Educate Pregnant Women about Prenatal Screening: A Randomized Controlled Study. Am J Perinatol. 2019 Feb;36(3):322-328. doi: 10.1055/s-0038-1667371. Epub 2018 Aug 14. PMID 30107621
- [Background] Kuppermann M, Pena S, Bishop JT, Nakagawa S, Gregorich SE, Sit A, Vargas J, Caughey AB, Sykes S, Pierce L, Norton ME. Effect of enhanced information, values clarification, and removal of financial barriers on use of prenatal genetic testing: a randomized clinical trial. JAMA. 2014 Sep 24;312(12):1210-7. doi: 10.1001/jama.2014.11479. PMID 25247517
- [Background] Yee LM, Wolf M, Mullen R, Bergeron AR, Cooper Bailey S, Levine R, Grobman WA. A randomized trial of a prenatal genetic testing interactive computerized information aid. Prenat Diagn. 2014 Jun;34(6):552-7. doi: 10.1002/pd.4347. Epub 2014 Mar 18. PMID 24578289
- [Background] Bryant AS, Norton ME, Nakagawa S, Bishop JT, Pena S, Gregorich SE, Kuppermann M. Variation in Women's Understanding of Prenatal Testing. Obstet Gynecol. 2015 Jun;125(6):1306-1312. doi: 10.1097/AOG.0000000000000843. PMID 26000501
- [Background] Khoshnood B, Pryde P, Wall S, Singh J, Mittendorf R, Lee KS. Ethnic differences in the impact of advanced maternal age on birth prevalence of Down syndrome. Am J Public Health. 2000 Nov;90(11):1778-81. doi: 10.2105/ajph.90.11.1778. PMID 11076250
- [Background] Bishop J, Huether CA, Torfs C, Lorey F, Deddens J. Epidemiologic study of Down syndrome in a racially diverse California population, 1989-1991. Am J Epidemiol. 1997 Jan 15;145(2):134-47. doi: 10.1093/oxfordjournals.aje.a009084. PMID 9006310
- [Background] Dormandy E, Michie S, Hooper R, Marteau TM. Low uptake of prenatal screening for Down syndrome in minority ethnic groups and socially deprived groups: a reflection of women's attitudes or a failure to facilitate informed choices? Int J Epidemiol. 2005 Apr;34(2):346-52. doi: 10.1093/ije/dyi021. Epub 2005 Feb 28. PMID 15737971

DOCUMENTS (1):
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT07077707/ICF_000.pdf